CLINICAL TRIAL: NCT04103099
Title: Evaluation of the Impact of the HLNatural, Inc. Immune Support Product in Reducing the Length of Cold Symptoms in Adults Suffering From the Common Cold
Brief Title: Impact of HLNatural Immune Supplement on Colds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hawthorne Effect Inc. (Other)
Collaborators: HLNatural, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00037635
Record Dates: First submitted 2019-09-13; First posted 2019-09-25 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Immune System Diseases
MeSH Terms: conditions — Immune System Diseases

STUDY DESIGN:
Intervention Model Description: The present study will be a single site, prospective, single arm observational study of minimal risk consisting of at least 200 participants who suffer from cold symptoms
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HLNatural Immune Cohort (Other): Observational one arm virtual study of HLNatural Immune supplement
  Interventions: Dietary Supplement: HLNatural Immune

INTERVENTIONS:
Dietary Supplement: HLNatural Immune — Vitamin C, Echinacea, Ivy Extract, Zinc, Ginger and Turmeric in a powder form mixed with water

SUMMARY:
According to the Centers of Disease Control and Prevention (CDC) adults will have an average of 2-3 colds per year. Most colds will last approximately 7-10 days. The symptoms of colds could include cough, sore throat, runny nose, body aches, fevers, headaches and fatigue. A cold can affect your activity such as going to work, interrupting your sleep and your day to day activities. The test product contains all natural ingredients which have been combined into a powder to be taken in water at the sign of a cold.

DETAILED DESCRIPTION:
At the onset of a cold, mix 1 packet of the drink-mix product in 6-8 oz. of hot water. Drink the drink mix twice a day until symptoms are gone or 18 days, whichever comes first.

1. Complete the screening survey.
2. Sign the eConsent if approved.
3. Complete the baseline survey, demographic form, and Medication and Supplements form.
4. Receive test product and log into study portal and complete supplement receipt form. This will mark the start of your participation in this study.
5. Once you have a cold, complete the symptom survey.
6. Take test product.
7. Write down any adverse or ill effects any time after taking the test product.
8. Record if you took any additional medications or supplements daily during the course of your cold.
9. Note any final adverse events and complete the exit form.

ELIGIBILITY:
Inclusion Criteria:

Adult candidates in the general population who are in good health and are seeking herbal remedies to reduce the duration of their common cold symptoms when they should arise. Participants will be deemed to be in good health if they do not report any of the medical conditions asked about in the screening questionnaire.

Exclusion Criteria:

* Age < 18 years old
* Unwilling to try the test product during their first cold experience in the trial
* Has any of the following medical conditions:

  * Chronic seasonal allergies
  * Allergy to any of the following ingredients: Echinacea, Ivy Extract, Camu Camu, Vitamin C, Ginger, Turmeric, Zinc or a known allergy to Guar Gum, Monk Fruit, Citric Acid, Natural Flavors.
  * Asthma
  * Current cold infection
  * Currently taking antimicrobial or antiviral medication
  * Alcohol consumption more than 7 drinks per week or more than 3 drinks per occasion
  * Routine recreational drug use
  * Chronic renal disease
  * Chronic liver disease
  * Known autoimmune or immunodeficiency disorders
  * Medically treated atopy or allergy
  * Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2019-10-16 (Actual); Primary Completion 2020-08-15 (Actual); Study Completion 2020-08-15 (Actual)

PRIMARY OUTCOMES:
Outcome of freedom of cold symptoms while consuming HLNatural Supplement | At the onset of cold symptoms the symptoms will be measured for 18 days or sooner if the symptoms resolve.
  Cold symptoms will be measured until the symptoms resolve. Subjects must experience 2 of more symptoms which are: cough, hoarseness, muscle aches, nasal drainage, nasal congestion, scratchy throat, sore throat, sneezing, or an oral temperature of 37.7 C (99.9 F).

SECONDARY OUTCOMES:
Outcome of the severity of cold symptoms while taking HLNatural Supplement | The diary will be completed daily during the duration of the the subject's cold.
  Subjects will rate the severity of the cold symptoms using Daily Symptom Survey of each possible symptom from 0-3 (3 is severe).
  * Comparison against the participant's normal behavior.
  * Net Promoter Score.
  * Adverse events will be summarized.
  * An additional data presentation will consist of results from both Treatment and Control in similar studies appearing in the literature. There will be no formal statistical comparison of results from this study and historical studies.
Outcome of the duration of the cold symptoms while taking HLNatural Supplement | At the onset of cold symptoms until resolution of cold symptoms
  The length of time that the subject's cold will be recorded
Required Behavior | During the duration of the cold symptoms
  Subjects will be asked to avoid over the counter cold-relief medication. However pain relievers and fever reducers are allowed
Outcome all adverse events while taking HLNatural Supplement | Throughout the study
  All adverse events which are collected throughout the subjects participation will be recorded.
Outcome of natural behavior of the participants while taking in the clinical trial | The subject will complete the screening, demographic and baseline surveys prior to the start of the product and the exit form at the end of the subject's cold symptoms
  All subjects will be asked to complete a screening, demographic and baseline questionnaire as well as and exit survey. The screening and baseline survey will be used to understand the subjects normal behavior with cold symptoms. The Exit study will rate the product to understand if the subject felt it helped with their cold symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Soynoa Rafatajah, MD, Principal Investigator — Hawthorne Effect Inc.
Locations (1):
- Hawthorne Effect, Inc., Lafayette, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abdollahi E, Momtazi AA, Johnston TP, Sahebkar A. Therapeutic effects of curcumin in inflammatory and immune-mediated diseases: A nature-made jack-of-all-trades? J Cell Physiol. 2018 Feb;233(2):830-848. doi: 10.1002/jcp.25778. Epub 2017 Mar 31. PMID 28059453
- [Background] Clinic, M. Vitamin C. 2017, October 18; Available from: https://www.mayoclinic.org/drugs-supplements-vitamin-c/art-20363932.
- [Background] Fazio S, Pouso J, Dolinsky D, Fernandez A, Hernandez M, Clavier G, Hecker M. Tolerance, safety and efficacy of Hedera helix extract in inflammatory bronchial diseases under clinical practice conditions: a prospective, open, multicentre postmarketing study in 9657 patients. Phytomedicine. 2009 Jan;16(1):17-24. doi: 10.1016/j.phymed.2006.05.003. Epub 2006 Jul 24. PMID 16860549
- [Background] Fonseca FN, Papanicolaou G, Lin H, Lau CB, Kennelly EJ, Cassileth BR, Cunningham-Rundles S. Echinacea purpurea (L.) Moench modulates human T-cell cytokine response. Int Immunopharmacol. 2014 Mar;19(1):94-102. doi: 10.1016/j.intimp.2013.12.019. Epub 2014 Jan 13. PMID 24434371
- [Background] Fulgoni VL 3rd, Keast DR, Bailey RL, Dwyer J. Foods, fortificants, and supplements: Where do Americans get their nutrients? J Nutr. 2011 Oct;141(10):1847-54. doi: 10.3945/jn.111.142257. Epub 2011 Aug 24. PMID 21865568
- [Background] Gammoh NZ, Rink L. Zinc in Infection and Inflammation. Nutrients. 2017 Jun 17;9(6):624. doi: 10.3390/nu9060624. PMID 28629136
- [Background] Grosso G, Bei R, Mistretta A, Marventano S, Calabrese G, Masuelli L, Giganti MG, Modesti A, Galvano F, Gazzolo D. Effects of vitamin C on health: a review of evidence. Front Biosci (Landmark Ed). 2013 Jun 1;18(3):1017-29. doi: 10.2741/4160. PMID 23747864
- [Background] Hemila H, Petrus EJ, Fitzgerald JT, Prasad A. Zinc acetate lozenges for treating the common cold: an individual patient data meta-analysis. Br J Clin Pharmacol. 2016 Nov;82(5):1393-1398. doi: 10.1111/bcp.13057. Epub 2016 Jul 28. PMID 27378206
- [Background] Hilding DA. Literature review: the common cold. Ear Nose Throat J. 1994 Sep;73(9):639-43, 46-7. PMID 7988393
- [Background] Hudson JB. Applications of the phytomedicine Echinacea purpurea (Purple Coneflower) in infectious diseases. J Biomed Biotechnol. 2012;2012:769896. doi: 10.1155/2012/769896. Epub 2011 Oct 26. PMID 22131823
- [Background] Jawad M, Schoop R, Suter A, Klein P, Eccles R. Safety and Efficacy Profile of Echinacea purpurea to Prevent Common Cold Episodes: A Randomized, Double-Blind, Placebo-Controlled Trial. Evid Based Complement Alternat Med. 2012;2012:841315. doi: 10.1155/2012/841315. Epub 2012 Sep 16. PMID 23024696
- [Background] Lang C, Rottger-Luer P, Staiger C. A Valuable Option for the Treatment of Respiratory Diseases: Review on the Clinical Evidence of the Ivy Leaves Dry Extract EA 575(R). Planta Med. 2015 Aug;81(12-13):968-74. doi: 10.1055/s-0035-1545879. Epub 2015 Apr 15. PMID 25875509
- [Background] Langley PC, Pergolizzi JV Jr, Taylor R Jr, Ridgway C. Antioxidant and associated capacities of Camu camu (Myrciaria dubia): a systematic review. J Altern Complement Med. 2015 Jan;21(1):8-14. doi: 10.1089/acm.2014.0130. Epub 2014 Oct 2. PMID 25275221
- [Background] Lopresti AL, Hood SD, Drummond PD. Multiple antidepressant potential modes of action of curcumin: a review of its anti-inflammatory, monoaminergic, antioxidant, immune-modulating and neuroprotective effects. J Psychopharmacol. 2012 Dec;26(12):1512-24. doi: 10.1177/0269881112458732. Epub 2012 Oct 3. PMID 23035031
- [Background] Matthias A, Banbury L, Stevenson LM, Bone KM, Leach DN, Lehmann RP. Alkylamides from echinacea modulate induced immune responses in macrophages. Immunol Invest. 2007;36(2):117-30. doi: 10.1080/08820130600745786. PMID 17365014
- [Background] Matthias A, Banbury L, Bone KM, Leach DN, Lehmann RP. Echinacea alkylamides modulate induced immune responses in T-cells. Fitoterapia. 2008 Jan;79(1):53-8. doi: 10.1016/j.fitote.2007.07.012. Epub 2007 Aug 11. PMID 17855021
- [Background] McMahon, G., Comparison of a Numeric and a Descriptive Pain Scale in the Occupational Medicine Setting. 2019.
- [Background] Trumbo P, Yates AA, Schlicker S, Poos M. Dietary reference intakes: vitamin A, vitamin K, arsenic, boron, chromium, copper, iodine, iron, manganese, molybdenum, nickel, silicon, vanadium, and zinc. J Am Diet Assoc. 2001 Mar;101(3):294-301. doi: 10.1016/S0002-8223(01)00078-5. No abstract available. PMID 11269606
- [Background] Mossad SB, Macknin ML, Medendorp SV, Mason P. Zinc gluconate lozenges for treating the common cold. A randomized, double-blind, placebo-controlled study. Ann Intern Med. 1996 Jul 15;125(2):81-8. doi: 10.7326/0003-4819-125-2-199607150-00001. PMID 8678384
- [Background] Mozaffari-Khosravi H, Naderi Z, Dehghan A, Nadjarzadeh A, Fallah Huseini H. Effect of Ginger Supplementation on Proinflammatory Cytokines in Older Patients with Osteoarthritis: Outcomes of a Randomized Controlled Clinical Trial. J Nutr Gerontol Geriatr. 2016 Jul-Sep;35(3):209-18. doi: 10.1080/21551197.2016.1206762. PMID 27559855
- [Background] Oregon State University, M.I.C. Zinc. Available from: https://lpi.oregonstate.edu/mic/minerals/zinc#reference175
- [Background] Project, R. The R Project for Statistical Computing.; Available from: https://www.R-project.org/.
- [Background] Rahnama P, Montazeri A, Huseini HF, Kianbakht S, Naseri M. Effect of Zingiber officinale R. rhizomes (ginger) on pain relief in primary dysmenorrhea: a placebo randomized trial. BMC Complement Altern Med. 2012 Jul 10;12:92. doi: 10.1186/1472-6882-12-92. PMID 22781186
- [Background] Raman, R., MS, RD. Echinacea: Benefits, Uses, Side Effects and Dosage. . 2018, October 15; Available from: https://www.healthline.com/nutrition/echinacea#side-effects.
- [Background] Sexton, D.M.M. The common cold in adults: Diagnosis and clinical features. 2018, February 22; Available from: https://www.uptodate.com/contents/the-common-cold-in-adults-diagnosis-and-clinical-features?csi=b9dba3ea-808c-423c-aa05-d1f3771bf7d5&source=contentShare.
- [Background] Shah SA, Sander S, White CM, Rinaldi M, Coleman CI. Evaluation of echinacea for the prevention and treatment of the common cold: a meta-analysis. Lancet Infect Dis. 2007 Jul;7(7):473-80. doi: 10.1016/S1473-3099(07)70160-3. PMID 17597571
- [Background] Sultan MT, Butt MS, Qayyum MM, Suleria HA. Immunity: plants as effective mediators. Crit Rev Food Sci Nutr. 2014;54(10):1298-308. doi: 10.1080/10408398.2011.633249. PMID 24564587
- [Background] Thamlikitkul L, Srimuninnimit V, Akewanlop C, Ithimakin S, Techawathanawanna S, Korphaisarn K, Chantharasamee J, Danchaivijitr P, Soparattanapaisarn N. Efficacy of ginger for prophylaxis of chemotherapy-induced nausea and vomiting in breast cancer patients receiving adriamycin-cyclophosphamide regimen: a randomized, double-blind, placebo-controlled, crossover study. Support Care Cancer. 2017 Feb;25(2):459-464. doi: 10.1007/s00520-016-3423-8. Epub 2016 Oct 6. PMID 27714530
- [Background] Van Straten M, Josling P. Preventing the common cold with a vitamin C supplement: a double-blind, placebo-controlled survey. Adv Ther. 2002 May-Jun;19(3):151-9. doi: 10.1007/BF02850271. PMID 12201356
- [Background] Wat D. The common cold: a review of the literature. Eur J Intern Med. 2004 Apr;15(2):79-88. doi: 10.1016/j.ejim.2004.01.006. PMID 15172021
- [Background] WebMD, English Ivy: Uses, Side Effects, Interactions, Dosage, and Warning
- [Background] WebMD. Ginger: Uses, Side Effects, Interactions, Dosage, and Warning.; Available from: https://www.webmd.com/vitamins/ai/ingredientmono-961/ginger.
- [Background] WebMD. Zinc: Uses, Side Effects, Interactions, Dosage, and Warning.; Available from: https://www.webmd.com/vitamins/ai/ingredientmono-982/zinc.
- [Background] Wessels I, Maywald M, Rink L. Zinc as a Gatekeeper of Immune Function. Nutrients. 2017 Nov 25;9(12):1286. doi: 10.3390/nu9121286. PMID 29186856
- [Background] Xu XY, Meng X, Li S, Gan RY, Li Y, Li HB. Bioactivity, Health Benefits, and Related Molecular Mechanisms of Curcumin: Current Progress, Challenges, and Perspectives. Nutrients. 2018 Oct 19;10(10):1553. doi: 10.3390/nu10101553. PMID 30347782
- [Background] Yale SH, Liu K. Echinacea purpurea therapy for the treatment of the common cold: a randomized, double-blind, placebo-controlled clinical trial. Arch Intern Med. 2004 Jun 14;164(11):1237-41. doi: 10.1001/archinte.164.11.1237. PMID 15197051
- [Background] Pappas, Diane E. Epidemiology, clinical manifestation, and pathogensis of rhinovirus infections. Available from: https://www.uptodate.com/contents/epidemiology-clinical-manifestations-and-pathogenesis-of-rhinovirus-infections?search=common%20cold%20cytokine&source=search_result&selectedTitle=1~150&usage_type=default&display_rank=1#H8
- [Background] Solomon, Daniel H. Non-selective NSAIDs: Overview of adverse effects. Available from: https://www.uptodate.com/contents/nonselective-nsaids-overview-of-adverse-effects?search=side%20effects%20of%20nsaids&source=search_result&selectedTitle=1~150&usage_type=default&display_rank=1#H22
- [Background] Lexicom, Inc. Phenylephrine (systemic): Drug Information. Available from: https://www.uptodate.com/contents/phenylephrine-systemic-drug-information?search=phenylephrine%20decongestant%20adult&source=search_result&selectedTitle=3~25&usage_type=default&display_rank=3#F9504784

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-07-17): https://cdn.clinicaltrials.gov/large-docs/99/NCT04103099/Prot_SAP_ICF_000.pdf